CLINICAL TRIAL: NCT02540447
Title: Graft Portal Reperfusion Without Purging Graft Preservative Solution In Living Donor Liver Transplantation. A Prospective Randomized Controlled Trial
Brief Title: Purge Vs no Purge in Living Donor Liver Transplantation Recipients
Acronym: PNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Yassen, Professor of Anesthesia and Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Purge_LTX
Record Dates: First submitted 2015-08-30; First posted 2015-09-04 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2016-12

CONDITIONS: Ischemia Reperfusion Injury
Keywords: Liver transplantation; Graft rinse; Ischemia reperfusion injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purge (Experimental): The donor surgical team excised the right liver lobe (without inclusion of the middle hepatic vein) and preserved it on the back table with cold custodiol (4°C solution, Portal vein (PV) was completely anastomosed and the right hepatic vein (RHV) was anastomosed with the recipient hepatic vein apart from last suture" that was left for drainage of the liver graft contents of the preservative solution into the peritoneal cavity using portal blood after portal declamping based on the graft volume and suctioned through an external sucker, then completed the RHV anastomosis.
  Interventions: Procedure: Purge
- No Purge (No Intervention): The donor surgical team excised the right liver lobe (without inclusion of the middle hepatic vein) and preserved it on the back table with cold Custodiol (4°C solution, Both portal vein and RHV were completely anastomosed prior to portal declamping and the graft preservative contents were washed into the systemic circulation by the portal blood at portal declamping.

INTERVENTIONS:
Procedure: Purge — In the recipient before portal declamping, the graft preservative solution and the mesenteric blood is washed out of the circulation into the abdominal cavity and sucked by external sucker through the incompletely anastomosed hepatic vein prior to portal declamping
  Arms: Purge

SUMMARY:
The investigators tested the impact of purging the graft contents and mesenteric blood into the systemic circulation versus washing out this volume out of the circulation in living donor liver transplantation recipients.

DETAILED DESCRIPTION:
All donors had right hepatectomy. On the back table, surgeons flushed liver grafts with 4 Liters of cold Custodiol solution. Patients were randomized into either purge group (Pg) (n=40) were graft fluid contents were washed out by the patient's portal vein blood (0.5ml per gram graft weight) through incompletely anastomosed hepatic vein, or No purge group (NPg) (n=40) where graft fluid contents were washed into the systemic circulation by the patient's portal blood. The primary outcome objective was the mean arterial blood pressure 5 minutes after portal declamping. Secondary objectives included hemodynamic and oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Adult living donor liver transplantation recipients of either sex in mansoura liver transplantation program

Exclusion Criteria:

* re-transplantation
* Previous upper abdominal operation
* Budd Chiari syndrome

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Yassen, MD, Principal Investigator — Mansoura Faculty of Medicine
Locations (1):
- Liver transplantation project - Gastroenterology surgical center - Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Candidates recruited from patients admitted for living donor liver transplantation in Mansoura liver transplantation unit
Groups:
- Purge: The donor surgical team excised the right liver lobe (without inclusion of the middle hepatic vein) and preserved it on the back table with cold custodiol (4°C solution, Portal vein (PV) was completely anastomosed and the right hepatic vein (RHV) was anastomosed with the recipient hepatic vein apart from last suture" that was left for drainage of the liver graft contents of the preservative solution into the peritoneal cavity using portal blood after portal declamping based on the graft volume and suctioned through an external sucker, then completed the RHV anastomosis.
  Purge of graft contents out of the circulation: In the recipient before portal declamping, the graft preservative solution and the mesenteric blood is washed out of the circulation into the abdominal cavity and sucked by external sucker through the incompletely anastomosed hepatic vein prior to portal declamping
Period: Overall Study
Arm/Group | Purge | No Purge
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Purge | No Purge | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (6.19) | 50.9 (7.62) | 51.15 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 32 | 34 | 66
Region of Enrollment [Number; unit: participants]
  Egypt | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Lowest 5 Minutes Post-reperfusion Mean Arterial Blood Pressure
Description: The lowest of three recorded mean arterial pressure readings at 1,3 and 5 minutes after portal declamping
Time Frame: 5 minutes post-reperfusion
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Purge: Portal vein (PV) was completely anastomosed and the right hepatic vein (RHV) was anastomosed with the recipient hepatic vein apart from last suture" that was left for drainage of the liver graft contents of the preservative solution into the peritoneal cavity using portal blood after portal declamping based on the graft volume and suctioned through an external sucker, then completed the RHV anastomosis.
  Purge of graft contents out of the circulation: In the recipient before portal declamping, the graft preservative solution and the mesenteric blood is washed out of the circulation into the abdominal cavity and sucked by external sucker through the incompletely anastomosed hepatic vein prior to portal declamping
- No Purge: Both portal vein and RHV were completely anastomosed prior to portal declamping and the graft preservative contents were washed into the systemic circulation by the portal blood at portal declamping.
Arm/Group | Purge | No Purge
Number analyzed (Participants) | 40 | 40
mmHg | 66.03 (6.13) | 57.75 (5.91)

2. Secondary Outcome: Biliary Complications (Participants)
Description: Participants who developed biliary complications in three months period (Participant)
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Purge | No Purge
Number analyzed (Participants) | 40 | 40
participants | 10 | 6

3. Secondary Outcome: Ischemia Reperfusion Injury
Description: incidence of ischemia reperfusion injury in the transplanted graft
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Purge | No Purge
Number analyzed (Participants) | 40 | 40
participants | 3 | 2

4. Secondary Outcome: Post-operative Infectious Complications
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Purge | No Purge
Number analyzed (Participants) | 40 | 40
participants | 9 | 8

5. Secondary Outcome: 3 Months Mortality
Description: mortality within first 3 post-operative months
Time Frame: 3 Months
Measure: Number; unit: participants
Arm/Group | Purge | No Purge
Number analyzed (Participants) | 40 | 40
participants | 4 | 3

ADVERSE EVENTS:
Time Frame: 3 months complications
Arm/Group | Purge | No Purge
Serious Adverse Events (participants affected / at risk) | 4/40 | 3/40
Other Adverse Events (participants affected / at risk) | 18/40 | 15/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Purge (N=40) | No Purge (N=40)
3 Months Mortality (Surgical and medical procedures) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Purge (N=40) | No Purge (N=40)
30 days morbidity (Surgical and medical procedures) | 18 (35) | 15 (34) — NonLife threatening complications including infection, acute cellular rejection, vascular complications, biliary complications and IR injury
Infectious complications (30 days) (Infections and infestations) | 5 (9) | 6 (8) — Early infectious complications
Acute cellular rejection (30 Days) (Immune system disorders) | 12 (12) | 15 (15)
Ischemia/Reperfusion Injury (30 days) (General disorders) | 3 (3) | 2 (2)
Billiary complications (30 Days) (Hepatobiliary disorders) | 10 (10) | 6 (6)
Vascular complications (30 Days) (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes